CLINICAL TRIAL: NCT02776618
Title: Aesthetic and Functional Efficacy of Poliglecaprone 25 vs Polyglactin 910 in Running Subcuticular Closures: a Split-scar, Rater-blinded Randomized Controlled Trial
Brief Title: Polyglactin 910 vs Poligelecaprone 25 Running Subcuticular Closure of Elliptical Excision Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: could not and did not recruit any participants
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Scott Worswick, Health Sciences Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #15-001216
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Cosmetics, Suture, Cicatrix
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyglactin 910 (Experimental): One half of excision site will be randomly assigned superficial closure with polyglactin 910 suture
  Interventions: Procedure: running subcuticular closure of excisional defect
- poliglecaprone 25 (Experimental): One half of excision site will be randomly assigned superficial closure with poliglecaprone 25
  Interventions: Procedure: running subcuticular closure of excisional defect

INTERVENTIONS:
Procedure: running subcuticular closure of excisional defect — Excisional defects will be repaired with deep polyglactin 910 sutures, followed by each half of the wound given randomly assigned subcuticular superficial closure as described in the treatment arms.

SUMMARY:
We will be recruiting patients requiring excisions of skin cancer and comparing aesthetic and functional differences of suture repair of excisional defects using polyglactin 910 vs poliglecaprone 25 with a split-scar model. Excision sites will be on either the trunk or extremities. Standard dermatological excision and repair methods will be used for removal of lesions and repair of the wound by surgeons; training courses will be used to limit inter-surgeon variation in technique. Excisional defects will be repaired with deep polyglactin 910 sutures, followed by randomly assigned subcuticular closure of one half of the defect with polyglactin 910 sutures and the other half with poliglecaprone 25 sutures. The patient will follow-up at 6 months and fill out a patient self-assessment evaluation survey of the scar. Photographs will also be taken of the scars at the follow-up at 6 months, which will be then be assigned to a set of blinded observers to evaluate the wound using a modified Patient Observer Self-Assessment Scale (mPOSAS). These observers will rate each scar on the mPOSAS scale and values will be averaged between observers. Total duration of participation will be 6 months, with 2 total visits (excision visit and follow-up visit).

DETAILED DESCRIPTION:
Screening: Patients will be recruited for the study after the need for excision of cutaneous malignancy has been been determined by biopsy. Patients who meet inclusion and exclusion criteria (please refer to section 11.1) will be offered to have an elliptical excision with repair by standard of care (surgeon's choice of closure of entire surgical wound) or be enrolled in the study. Patients will be recruited directly by the PI and/or co-investigators, typically on the telephone when biopsy results of cutaneous malignancy and the need for treatment by excision are being conveyed. Occasionally the patient's may be recruited directly in-person if a subsequent office-visit occurs between the patient and the physician. Patient's who enroll in the study will then undergo intervention with excision and repair at a time convenient to them, ideally within one month.

Intervention:

Patients will undergo a medically-necessary elliptical excision of their cutaneous malignancy using standard excision protocol. This will occur in a similar time frame to a standard excision of cutaneous malignancy in our clinics ranging from 1-4 weeks from diagnosis, based on the patient's preference and schedule. The wound will be divided into halves designated as side A (either left or superior aspect) and side B (either right or inferior). Side A of the wound will be randomly assigned subcuticular closure with either poliglecaprone 25 or polyglactin 910. Side B will receive the opposite of side A. Randomization will be performed with online randomization software (https://www.randomizer.org). Prior to placement of the superficial subcuticular sutures, both sides of the wound will receive vertical deep sub-epidermal sutures using polyglactin 910. Patients will be blinded as to which material is used on which side. After the wound is closed, a de-identified photograph will be taken by the PI or co-investigators of the wound with demarcation of sites A and B (using a surgical pen) to serve as a marker for side A and side B for future identification of the intervention sites. The type of randomized intervention to site A and site B will be recorded without identifying patient information on a secure, encrypted database. Closed wounds will be treated with standard protocol with a pressure bandage left in place for 24 hours followed by daily treatment with petrolatum ointment and a bandage for 2 weeks until the epidermis has healed together completely. Patients will be counseled on standard wound care as well as common complications of standard excisions by the surgeon. No visit for suture removal will be necessary as all sutures are dissolvable.

*note - interventional methods for patients included in the study are considered standard therapy. Patient's would still receive similar excision and closure of their wound if they were not participating in the research.

Follow-up:

Patients will be called via telephone by either the PI or co-investigators after 2 weeks to inquire about the healing process and assess for any complications.

Patients will then follow up at 6 months for their scheduled routine skin cancer surveillance exam with the surgeon who performed the excision. At that time, the surgeon will re-identify sites A and B with a surgical marking pen. A de-photograph will be taken of the excision site scar. At the end of the patient visit, the patient will personally given a POSAS patient survey and asked to rate their scar for both sites A and B; no identifying information will be included in this survey. In the case that the scar is in a location that the patient can not easily visualize, the de-identified photograph of the patient's scar will be printed for the patient to assess the scar. Photographs will then later be assigned to two blinded observers to assign a modified observer POSAS score to subjects' scars. These scores will be averaged and then analyzed for differences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older requiring excision of either cutaneous squamous cell carcinoma or basal cell carcinoma with postoperative defects of at least 4 cm on the trunk and extremities resulting from simple excisional defects. Participants will be patients of the dermatology departments of either the University of California, Los Angeles

Exclusion Criteria:

* pregnancy, incarceration, mental impairment, inability to understand English, nonlinear closures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Modified Patient and Observer Scar Assessment Scale | 6 month after surgery
  The Patient and Observer Scar Assessment Scale includes subjective symptoms of pain and pruritus and consists of 2 numerical numeric scales: The Patient Scar Assessment Scale and the Observer Scar Assessment Scale. It assesses vascularity, pigmentation, thickness, relief, pliability, and surface area, and it incorporates patient assessments of pain, itching, color, stiffness, thickness, and relief.

SECONDARY OUTCOMES:
Visual analog scale | 6 months after surgery
  The multidimensional visual analog scale is a photograph-based scale derived from evaluating standardized digital photographs in 4 dimensions (pigmentation, vascularity, acceptability, and observer comfort) plus contour.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Worswick, MD, Principal Investigator — Univeristy of California, Los Angeles
Locations (1):
- Department of Dermatology, University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No